CLINICAL TRIAL: NCT07149597
Title: Clinical Validation Study on the Imaging Efficacy of Mobile 4D CBCT Technology for Peripheral Pulmonary Lesions
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Director, Department of Respiratory Endoscopy, Shanghai Chest Hospital
Other Study IDs: IS25179
Record Dates: First submitted 2025-08-22; First posted 2025-09-02 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Peripheral Pulmonary Lesions (PPLs)
Keywords: Mobile Cone-Beam Computed Tomography; Artificial Intelligence; Peripheral Pulmonary Lesions

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mobile CBCT Group: This study aims to explore the clinical value of mobile 4D CBCT technology in the diagnosis and treatment of peripheral pulmonary lesions, and to validate its intraoperative three-dimensional CT imaging capability. Preoperative fluoroscopic localization will be performed, followed by two rounds of three-dimensional scanning using a mobile C-arm system to acquire volumetric CT images of the patients. The obtained images will be exported and processed postoperatively, and analyzed from both quantitative and qualitative perspectives.
  Interventions: Radiation: Mobile CBCT Three-Dimensional Scanning

INTERVENTIONS:
Radiation: Mobile CBCT Three-Dimensional Scanning — Mobile CBCT Three-Dimensional Scanning

SUMMARY:
The purpose of this study is to evaluate the clinical value of mobile 4D CBCT technology in the diagnosis and treatment of peripheral pulmonary lesions and to validate its intraoperative dynamic three-dimensional CT imaging capability.

DETAILED DESCRIPTION:
This is a single-arm, single-center, prospective study in which approximately 50 patients with peripheral pulmonary lesions will undergo mobile cone-beam computed tomography (CBCT) scanning. In the field of respiratory intervention, mobile CBCT enables real-time intraoperative three-dimensional CT imaging of lesions, providing a more intuitive visualization of the positional relationship between biopsy tools and the target area, offering significant value in bronchoscopic examinations. In this study, CBCT images will be acquired from participants and reconstructed into three-dimensional models. Subsequent analysis will be conducted to evaluate the performance of mobile 4D CBCT three-dimensional reconstruction technology.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years old.
2. Patients whose chest CT scans indicate the presence of peripheral pulmonary lesions and require further diagnosis via transbronchial lung biopsy (TBLB).
3. Lesion size: 8 mm < longest diameter of lesion ≤ 50 mm.
4. Understands the study and has provided signed informed consent.

Exclusion Criteria:

1. Contraindications to bronchoscopy are present.
2. Severe cardiopulmonary dysfunction or other conditions that may increase surgical risk.
3. The investigator considers that the patient has other conditions which make them unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent mobile CBCT scanning.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
RMSE（Root Mean Squared Error） | 1 year
  RMSE (Root Mean Square Error): A commonly used metric for measuring the difference between predicted values and actual values. It is applicable in regression problems and image quality assessment. A smaller RMSE value indicates more accurate predictions, with 0 representing perfect accuracy, while a larger value indicates greater error.
SSIM (Structural Similarity ) | 1 year
  SSIM (Structural Similarity ): A metric used to measure the similarity between two images, comparing them across three dimensions: luminance, contrast, and structure. The SSIM value ranges from [-1, 1], where 1 indicates that the two images are identical, and 0 or negative values indicate complete dissimilarity.

SECONDARY OUTCOMES:
Image Quality | 1 year
  Three experienced experts scored the three-dimensional CT reconstruction images based on image quality using the following criteria:4 points: Exceptionally clear images;3 points: Generally clear images with a few blurred slices;2 points: Basically clear images but with several blurred slices;1 point: Unclear images.
Slice Continuity | 1 year
  Three experienced experts scored the three-dimensional CT reconstruction images based on slice continuity using the following criteria:4 points: All slices exhibit continuous anatomical structures;3 points: Overall continuous with minor discontinuities in a few slices;2 points: Generally continuous but with noticeable discontinuities in multiple slices;1 point: Predominantly discontinuous across most slices.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, Study Director — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No